CLINICAL TRIAL: NCT03585153
Title: Multicenter Assessment of the Pancreas in Type 1 Diabetes
Acronym: MAP-T1D
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Texas at Austin (Other); University of Chicago (Other); University of Colorado, Denver (Other); St Vincent's Institute of Medical Research (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Daniel Moore, Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 130883; 3-SRA-2019-759-M-B (Other Grant/Funding Number: JDRF); 3-SRA-2015-102-M-B (Other Grant/Funding Number: JDRF)
Record Dates: First submitted 2018-06-18; First posted 2018-07-12 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood; mouth saliva swab; urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Individuals with stage 3 T1D: Individuals with overt stage 3 type 1 diabetes
  Interventions: Other: Non-contrast magnetic resonance imaging
- Healthy control: Individuals without type 1 diabetes
  Interventions: Other: Non-contrast magnetic resonance imaging
- Autoantibody positive: Individuals with early stage type 1 diabetes (stage 1, stage 2) who possess two or more type 1 diabetes-related autoantibodies
  Interventions: Other: Non-contrast magnetic resonance imaging
- Monogenic diabetes: Individuals with monogenic diabetes
  Interventions: Other: Non-contrast magnetic resonance imaging

INTERVENTIONS:
Other: Non-contrast magnetic resonance imaging — subjects lie in an MRI machine (non-contrast) for 30 minutes while we take pictures of their pancreas

SUMMARY:
The overall goal of this research is to develop and validate standard operating procedures (SOP) to assess the human pancreas in individuals with type 1 diabetes (T1D) and other forms of diabetes using advanced, quantitative magnetic resonance imaging (MRI) approaches.

DETAILED DESCRIPTION:
This research applies magnetic resonance imaging (MRI) techniques to study the pancreas of individuals with type 1 diabetes (T1D) and other forms of diabetes. Recent studies have demonstrated reduced pancreatic volume is present within months of T1D diagnosis in children, adolescents, and adults, and in non-diabetic individuals expressing islet autoantibodies that portend the development of T1D. As the pancreatic beta cells constitute only 1-2% of the pancreas, the degree of reduction in pancreas volume at disease onset suggests exocrine involvement, challenging the established paradigm of T1D being solely a disease of the endocrine pancreas. These unexpected findings raise fundamental questions that challenge our understanding of T1D pathogenesis. These changes in pancreatic volume and size before and soon after onset of T1D, as detected by MRI, appear to be a marker of the T1D pathogenic disease process. There is an urgent need to determine whether similar observations can be obtained at different centers using different MRI platforms. Discovery of unknown changes may lead to new ways to treat disease. The MRI techniques may also be useful for following how T1D is progressing in different people, determining whether new drugs are effective, and ultimately detecting T1D in people earlier than currently possible.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 8 years of age
* Subjects with T1D must be imaged within 100 days of their date of diagnosis
* Subjects must be able to read and provide assent/informed written consent

Exclusion Criteria:

* Subjects with pancreatitis, cystic fibrosis, pancreatic adenocarcinoma, or neuroendocrine tumors
* Subjects who have any type of bioimplant activated by mechanical, electronic, or magnetic means because such devices may be displaced or malfunction
* Subjects who have any type of ferromagnetic bioimplant that could potentially be displaced
* Subjects who are pregnant or breast-feeding. Urine pregnancy test will be performed on women of child bearing potential who are not practicing appropriate contraception measures or menstruating.
* Subjects who exhibit significant anxiety and/or claustrophobia
* Subjects incapable of giving assent/informed written consent
* For controls: subjects who have first degree relatives with T1D

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with diabetes for this study may be referred by any pediatric or adult endocrinologists. Healthy controls are recruited via a passive recruitment process. A small subset of controls will travel to multiple study centers to have an MRI. In this study, the MRI scan will be used for research purposes only. However, if we see something that is not normal, the participant will be told and asked to consult his or her doctor.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-02-19 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Pancreas Volume Index | up to 10 years
  Size of the pancreas determined by longitudinal MRI, normalized to subject weight

SECONDARY OUTCOMES:
MRI of pancreas - Apparent Diffusion Coefficient | up to 10 years
  MRI texture of pancreas

CONTACTS AND LOCATIONS:
Overall Officials: Alvin C. Powers, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (5):
- United States (4):
  - University of Colorado, Barbara Davis Center, Aurora, Colorado
  - University of Chicago, Kovler Diabetes Center, Chicago, Illinois
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas at Austin, Dell Medical School, Austin, Texas
- St. Vincent's Institute of Medical Research, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Virostko J, Williams J, Hilmes M, Bowman C, Wright JJ, Du L, Kang H, Russell WE, Powers AC, Moore DJ. Pancreas Volume Declines During the First Year After Diagnosis of Type 1 Diabetes and Exhibits Altered Diffusion at Disease Onset. Diabetes Care. 2019 Feb;42(2):248-257. doi: 10.2337/dc18-1507. Epub 2018 Dec 14. PMID 30552135
- [Result] Williams JM, Hilmes MA, Archer B, Dulaney A, Du L, Kang H, Russell WE, Powers AC, Moore DJ, Virostko J. Repeatability and Reproducibility of Pancreas Volume Measurements Using MRI. Sci Rep. 2020 Mar 16;10(1):4767. doi: 10.1038/s41598-020-61759-9. PMID 32179809
- [Derived] Wright JJ, Dulaney A, Williams JM, Hilmes MA, Du L, Kang H, Powers AC, Moore DJ, Virostko J. Longitudinal MRI Shows Progressive Decline in Pancreas Size and Altered Pancreas Shape in Type 1 Diabetes. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2699-2707. doi: 10.1210/clinem/dgad150. PMID 36938587

DOCUMENTS (1):
  • Informed Consent Form (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03585153/ICF_000.pdf